CLINICAL TRIAL: NCT01405638
Title: Faith-based Approaches to Treating Hypertension and Colon Cancer Prevention
Acronym: FAITH-CRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 10-00427; 1R01HL096946-01A2 (NIH)
Record Dates: First submitted 2011-07-27; First posted 2011-07-29 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Blood Pressure; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Motivational Interviewing; Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Motivational Interviewing (Experimental): The use of a one-on-one motivational interviewing counseling intervention, 4 visits over 5 months, focusing on changes to behavior related to blood pressure control.
  Interventions: Behavioral: Motivational Interviewing
- Patient Navigation (Experimental): The use of a patient navigation intervention to guide participants through the process of getting screened for colorectal cancer.
  Interventions: Behavioral: Patient Navigation
- PLUS (Experimental): This group receives both the motivational interviewing intervention and the patient navigation intervention.
  Interventions: Behavioral: Motivational Interviewing; Behavioral: Patient Navigation

INTERVENTIONS:
Behavioral: Motivational Interviewing — One-on-one client-centered counseling for lifestyle changes related to blood pressure control
  Arms: Motivational Interviewing; PLUS
Behavioral: Patient Navigation — One-on-one navigation to guide participants through the process of being screened for colorectal cancer.
  Arms: PLUS; Patient Navigation

SUMMARY:
Primary Aim: To evaluate the effect of a lifestyle intervention delivered through telephone-based motivational interviewing (MINT) versus a patient navigation intervention on blood pressure reduction and CRC screening.

Hypotheses: Among black men, aged > 50 years with uncontrolled HTN and in need of CRC screening:

1. Hyp. 1: those randomized to the lifestyle intervention will have lower BP compared to those randomized to the patient navigation intervention at 6 months.
2. Hyp. 2: those randomized to the patient navigation intervention will have higher CRC screening rates compared to those randomized to the lifestyle intervention at 6 months.

DETAILED DESCRIPTION:
The primary outcomes will be (1) within-patient change in systolic and diastolic BP from baseline to 6 months and (2) CRC screening rates as determined by colonoscopy report or fecal immunochemical test (FIT) result from the primary care provider at 6 months. Blood pressure will be assessed with an automated digital BP monitor based on American Heart Association guidelines.1 CRC screening will be assessed by self-report and verified with medical records and/or the actual colonoscopy or FIT report from participants' providers.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be age 50 years or older
* Participants must have a working telephone (a necessary criterion since much of the interventions are telephone based)
* Self-identified as a black or African American and male
* Have uncontrolled hypertension defined as SBP>135 mmHg or DBP>85 mmHg and SBP >130 mmHg or DBP >80 mmHg (in those with diabetes) at the screening
* Have a need for CRC screening defined as: 1) no colonoscopy in the last 10 years; 2) no Flexible sigmoidoscopy, Digital Contrast Barium Enema or CT-colonoscopy in the last 5 years, or 3) no Fecal Immunochemical Test or Fecal Occult Blood Test in the last 12 months.
* All participants must be fluent in English. Certain measures used have not been verified in other languages.

Exclusion Criteria:

* Inability to comply with the study protocol (either self-selected or by indicating during screening that he could not complete all requested tasks).

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2011-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 6-months
  The primary outcomes will be (1) within-patient change in systolic and diastolic BP from baseline to 6 months and (2) CRC screening rates as determined by colonoscopy report or fecal immunochemical test (FIT) result from the primary care provider at 6 months. Blood pressure will be assessed with an automated digital BP monitor based on American Heart Association guidelines.1 CRC screening will be assessed by self-report and verified with medical records and/or the actual colonoscopy or FIT report from participants' providers.
Colorectal Cancer Screening | 6M
  The primary outcomes will be (1) within-patient change in systolic and diastolic BP from baseline to 6 months and (2) CRC screening rates as determined by colonoscopy report or fecal immunochemical test (FIT) result from the primary care provider at 6 months. Blood pressure will be assessed with an automated digital BP monitor based on American Heart Association guidelines.1 CRC screening will be assessed by self-report and verified with medical records and/or the actual colonoscopy or FIT report from participants' providers.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Ravenell, MD, MS, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States